CLINICAL TRIAL: NCT04367987
Title: Variability of Heart Rate as a Marker of Complication of Colorectal Surgery
Acronym: VFC COLORECTAL
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: Local/2018/MB-01
Record Dates: First submitted 2020-04-27; First posted 2020-04-29 (Actual); Last update posted 2022-03-21 (Actual); Status verified 2021-08

CONDITIONS: Surgery--Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients undergoing colorectal surgery
  Interventions: Diagnostic Test: Heart Rate Variability

INTERVENTIONS:
Diagnostic Test: Heart Rate Variability — Heart rate and RR interval Post-anonymized analysis of heart rate variability using the KUBIOS software

SUMMARY:
Heart rate variability reflects the autonomic nervous system on the intrinsic activity of sinus node cells. Sympathetic hyperactivity is an adaptation to stress, while parasympathetic hyperactivity is present at rest. Thus, any variability in the heart frequency rate reflects variations in sympathetic and parasympathetic components in the autonomic nervous system. Failure to return to normal or a reduction in the variability of the heart rate in the postoperative period is correlated with complications in colorectal surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients operated for a scheduled colorectal resection due to cancer, diverticulitis, or Chronic Inflammatory Bowel Disease,
* American Society of Anesthesiologists score 1-2
* The patient must have given their free and informed consent and signed the consent form
* The patient must be a member or beneficiary of a health insurance plan

Exclusion Criteria:

* Patient taking antidepressants, antipsychotics, antihypertensive beta blocker type, anti-arythmic or oral contraception
* Uncontrolled diabetes or associated with a neuropathy
* Arrhythmias and conduction disturbances, , coronaropathy and heart failure, kidney failure
* Neuropathies
* Pacemaker or defibrillator
* The subject is participating in another interventional study, or is in a period of exclusion determined by a previous study
* The subject refuses to sign the consent
* It is impossible to give the subject informed information
* The patient is under safeguard of justice or state guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients undergoing scheduled colorectal resection or operated on in the digestive surgery department of the CHU Nîmes
Sampling Method: Non-Probability Sample
Enrollment: 117 (Estimated)
Dates: Start 2020-06-17 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Rate of variability of the heart rate between Day-1 to Day 7 | Day 7
  Measured by power spectral density; ratio of the high to low frequencies
Correlation between the rate of variability of the heart rate between Day-1 to Day 7and anastomotic fistula diagnosed according to Center for Diseases Control criteria after scheduled colorectal surgery | Hospital discharge (maximum Day 7)
  Abdominal-pelvic imagery
Correlation between the rate of variability of the heart rate between Day-1 to Day 7 and peri-anastomotic fluid collections after scheduled colorectal surgery | Hospital discharge (maximum Day 7)
  Abdominal-pelvic imagery

SECONDARY OUTCOMES:
Correlation between the rate of variability of the heart rate between Day-1 to Day 7 and presence of intra abdominal abscess | Hospital discharge (maximum Day 7)
  diagnosed on CT-scan
Correlation between the rate of variability of the heart rate between Day-1 to Day 7 and presence of gut wall abscess | Hospital discharge (maximum Day 7)
Correlation between the rate of variability of the heart rate between Day-1 to Day 7 and presence of pneumonia | Hospital discharge (maximum Day 7)
Correlation between the rate of variability of the heart rate between Day-1 to Day 7 and presence of urinary tract infection | Hospital discharge (maximum Day 7)
Correlation between the rate of variability of the heart rate between Day-1 to Day 7 and presence of central venous catheter infection | Hospital discharge (maximum Day 7)
Correlation between the rate of variability of the heart rate between Day-1 to Day 7 and presence of intra abdominal hematoma | Hospital discharge (maximum Day 7)
Correlation between the rate of variability of the heart rate between Day-1 to Day 7 and presence of hemorrhagic shock | Hospital discharge (maximum Day 7)
Correlation between the rate of variability of the heart rate between Day-1 to Day 7 and death rate | Hospital discharge (maximum Day 7)
Correlation between the rate of variability of the heart rate between Day-1 to Day 7 and presence of deep vein thrombosis | Hospital discharge (maximum Day 7)
Correlation between the rate of variability of the heart rate between Day-1 to Day 7 and presence of pulmonary embolism | Hospital discharge (maximum Day 7)
Correlation between the rate of variability of the heart rate between Day-1 to Day 7 and presence of acute pulmonary edema | Hospital discharge (maximum Day 7)
Correlation between the rate of variability of the heart rate between Day-1 to Day 7 and presence of heart disease | Hospital discharge (maximum Day 7)

CONTACTS AND LOCATIONS:
Overall Officials: Martin Bertrand, Principal Investigator — CHU Nimes
Locations (1):
- CHU de Nimes, Nîmes, France